CLINICAL TRIAL: NCT05353413
Title: Diffusion Weighted Magnetic Resonance Imaging and the Optic Nerve Neuropathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Collaborators: University of Bialystok (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: R-I-002/477/2019
Record Dates: First submitted 2022-03-16; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-03

CONDITIONS: Ischemic Optic Neuropathy; Optic Neuritis; Compressive Optic Neuropathy; Traumatic Optic Neuropathy; Toxic Optic Neuropathy; Hereditary Optic Neuropathies
Keywords: optic neuropathies; visual evoked potential
MeSH Terms: conditions — Optic Neuropathy, Ischemic; Optic Neuritis; Optic Nerve Injuries; Toxic Optic Neuropathy; Optic Nerve Diseases | interventions — Neuroimaging

STUDY DESIGN:
Intervention Model Description: Two groups: volunteers with neuropathies and healthy volunteers
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Various types of optic neuropathies (Experimental): Patients with various types of optic neuropathy.
  Interventions: Device: Neuroimaging; Diagnostic Test: VEP - visual evoked potential; Diagnostic Test: Ophthalmology examination.
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Device: Neuroimaging; Diagnostic Test: VEP - visual evoked potential; Diagnostic Test: Ophthalmology examination.

INTERVENTIONS:
Device: Neuroimaging — Magnetic resonance diffusion tensor imaging of the brain
Diagnostic Test: VEP - visual evoked potential — Electrophysiology of the visual pathway.
Diagnostic Test: Ophthalmology examination. — Full ophthalmological examination (visual acuity, color vision, measurement of intraocular pressure, evaluation of the anterior chamber and the fundus of the eye using a slit lamp and the Volk lens, optical coherence tomography examination of the macula and optic nerve disc (OCT), neurological field vision)

SUMMARY:
The aim of the project is to create a new, non-invasive and safe protocol for the early diagnosis of various types of optic neuropathies with the use of diffusion magnetic resonance imaging

DETAILED DESCRIPTION:
In this study, it is planned to find twenty volunteers for each of the neuropathies and twenty healthy volunteers. Each volunteer will undergo clinical tests such as visual acuity, color vision, intraocular pressure measurement, assessment of the anterior chamber and fundus using a slit lamp and Volk lens, macular optical coherence tomography examination and examination of the optic nerve disc (OCT), neurological field vision and visual evoked potential (VEP) testing. Each of the volunteers will undergo magnetic resonance imaging. During active scanning, patients will be asked for not blinking or moving their heads by staring at the red dot on the outside of the camera reflected in the coil mirror. The obtained diffusion tensor data will be used for further analysis.

ELIGIBILITY:
Inclusion Criteria:

Optic neuropathy.

Exclusion Criteria:

common contraindications to MRI (presence of pacemaker, non-MRI-safety or claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
sigma parameter | one month
  sigma parameter in our algorithm provides a quantitative measure of nerve atrophy

CONTACTS AND LOCATIONS:
Locations (1):
- Lisowski, Wasilków, Poland

IPD SHARING:
Plan to Share IPD: No